CLINICAL TRIAL: NCT04711135
Title: A Multicenter Open-label Study to Evaluate Safety and Dosimetry of Lutathera in Adolescent Patients With Somatostatin Receptor Positive Gastroenteropancreatic Neuroendocrine (GEP-NET) Tumors, Pheochromocytoma and Paragangliomas (PPGL)
Brief Title: Study to Evaluate Safety and Dosimetry of Lutathera in Adolescent Patients With GEP-NETs and PPGLs
Acronym: NETTER-P
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAA601A32201; 2020-002951-39 (EudraCT Number); EMEA-002950-PIP01-20 (Other: EMA paediatric Investigation plan number(s) (PIP)); 2023-507444-37-00 (Other: EU CTIS)
Record Dates: First submitted 2020-12-16; First posted 2021-01-15 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumors; Pheochromocytoma; Paraganglioma
Keywords: GEP-NET; PPGL; adolescents; pediatric; Lutathera; Lutetium [177Lu] oxodotreotide; Lutetium Lu 177 dotatate; Peptide Receptor Radionuclide Therapy; PRRT
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Gastro-enteropancreatic neuroendocrine tumor | interventions — Lutetium; Lutetium-177; copper dotatate CU-64; lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GEP-NET and PPGL (Experimental): All eligible participants will receive Lutathera (7.4 GBq/200 mCi x 4 administrations every 8 weeks; cumulative dose: 29.6 GBq/800 mCi), with a concomitant administration of 2.5% Lysine - Arginine amino acid solution.
  Interventions: Drug: Lutetium [177Lu] oxodotreotide/dotatate

INTERVENTIONS:
Drug: Lutetium [177Lu] oxodotreotide/dotatate — Radiopharmaceutical solution for infusion (7.4 GBq of Lutathera per 30 ml vial)
  Other Names: Lutathera

SUMMARY:
This is a multicenter, open-label, single-arm study to evaluate the safety and dosimetry of Lutathera in adolescent patients 12 to <18 years old with somatostatin receptor positive GEP-NETs and PPGLs. The study will enroll at least 8 patients in the GEP-NET cohort and as many adolescents with PPGL as possible in the exploratory PPGL cohort.

DETAILED DESCRIPTION:
The study schedule for each patient consists of the screening period (up to 2 weeks) followed by the treatment period (4 treatment administrations at 8-week interval), and the follow-up period (10 years).

The treatment period will consist of 4 Lutathera treatments administered at 8-week intervals. Lutathera administration will occur on Week 1 Day 1 of each cycle. Each patient will receive a total of 4 doses of Lutathera (7.4 GBq/200 mCi x 4 administrations every 8 weeks; cumulative dose: 29.6 GBq/800 mCi). An infusion of 2.5% Lysine - Arginine amino acid (AA) solution will be co-administered with each Lutathera dose for renal protection according to the approved Lutathera local prescribing information. An antiemetic will be administered prior to infusion of the AA solution for prevention of infusion-related nausea and vomiting.

The dosimetry and PK assessments will be performed during the first week after the 1st Lutathera dose, i.e. one time during the study treatment period for each patient. The dosimetry analysis will allow for estimation from the 1st Lutathera administration of the cumulative absorbed radiation dose from 4 Lutathera doses and also for taking a decision on the next dose levels. In the exceptional circumstances when dosimetry cannot be performed in a particular patient after the first Lutathera dose, it should be completed as soon as feasible upon a later dose. In order to minimize risk for each study subject, an accelerated analysis of dosimetry and safety data will be performed for each patient in the study, to enable the Investigator to take a decision for the subsequent Lutathera doses. The results of dosimetry assessments (imaging and blood dosimetry) will be provided to the investigators for their evaluation prior to administration of subsequent therapeutic cycles in each patient.

A total follow-up period of 10 years (120 months) after the last Lutathera dose will take place for each patient who received at least one dose of Lutathera. This follow-up period will be comprised of a short-term follow-up of 6 months to evaluate cumulative Lutathera toxicities, followed by a long-term follow up of another 114 months.

An external Data and Safety Monitoring Board (DSMB) will also operate in the study to evaluate accumulating safety and dosimetry data, to ensure the safety of adolescents enrolled in the study, and to provide recommendations to investigators as well as to the clinical team in charge of conducting the study.

ELIGIBILITY:
Key Inclusion Criteria:

1. GEP-NET cohort: presence of metastasized or locally advanced, inoperable (curative intent), histologically proven, G1 or G2 (Ki-67 index =< 20%), well differentiated GEP-NET.

   or PPGL cohort: presence of metastasized or locally advanced, inoperable (curative intent), histologically proven PPGL.
2. Patients from 12 to < 18 years of age at the time of enrollment.
3. Expression of somatostatin receptors confirmed by a somatostatin receptor imaging (SRI) modality within 3 months prior to enrollment, with tumor uptake observed in the target lesions more or equal to the normal liver uptake.
4. Performance status as determined by Karnofsky score >= 50 or Lansky Play-Performance Scale score >= 50.
5. Parent's ability to understand and the willingness to sign a written informed consent document for adolescents as determined by local regulations. Adolescents will sign assent along with parental/legal guardian consent or will co-sign consent with parent/legal guardian in accordance with local regulation, prior to participation in the study.

Key Exclusion Criteria:

1. Laboratory parameters:

   1. Estimated creatinine clearance calculated by the Cockroft-Gault method < 70 mL/min
   2. Hb concentration <5.0 mmol/L (<8.0 g/dL); WBC <2x109/L; platelets <75x109/L.
   3. Total bilirubin >3 x ULN for age.
   4. Serum albumin <3.0 g/dL unless prothrombin time is within the normal range.
2. Established or suspected pregnancy.
3. Breastfeeding female patients unless they accept to discontinue breastfeeding from the 1st dose until 3 months after the last administration of study drug.
4. Female patients of child-bearing potential, unless they are using highly effective methods of contraception during treatment and for 6 months after the last dose of Lutathera.
5. Sexually active male patients, unless they agree to remain abstinent or be willing to use effective methods of contraception.
6. Patients for whom in the opinion of the investigator other therapeutic options are considered more appropriate than the therapy offered in the study, based on patient and disease characteristics.
7. Current spontaneous urinary incontinence.
8. Other known co-existing malignancies except non-melanoma skin cancer and carcinoma in situ of the uterine cervix, unless definitively treated and proven no evidence of recurrence for 5 years.
9. Hypersensitivity to the study drug active substance or to any of the excipients.
10. Patients with any other significant medical, psychiatric, or surgical condition, currently uncontrolled by treatment, which may interfere with the completion of the study.
11. Patient with known incompatibility to CT Scans with I.V. contrast due to allergic reaction or renal insufficiency. If such a patient can be imaged with MRI, then the patient would not be excluded.
12. Patients who received any investigational agent within the last 30 days.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2034-02-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (3):
  - University of Kentucky, Lexington, Kentucky
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Centre Léon Berard, Lyon, France
- Maria Sklodowska-Curie National Research Institute of Oncology, Gliwice, Poland
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- University College Hospital of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Gaze MN, Handkiewicz-Junak D, Hladun R, Laetsch TW, Sorge C, Sparks R, Wan S, Ceraulo A, Kluczewska-Galka A, Gamez-Cenzano C, States LJ, El Khouli R, Aimone P, Perraud K, Kollar G, Khanshan F, Blumenstein L, Brouri F, Giraudet AL. Safety and dosimetry of [177Lu]Lu-DOTA-TATE in adolescent patients with somatostatin receptor-positive gastroenteropancreatic neuroendocrine tumours, or pheochromocytomas and paragangliomas: Primary analysis of the Phase II NETTER-P study. Eur J Nucl Med Mol Imaging. 2025 Sep;52(11):4001-4015. doi: 10.1007/s00259-025-07246-7. Epub 2025 Apr 8. PMID 40198358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the data cut-off (DCO) date (12-Mar-2024) for this primary analysis 11 participants were enrolled across 7 centers.
Pre-assignment Details: The study schedule for each participant consisted of the screening period (up to 2 weeks) followed by the treatment period and the follow-up period.
Groups:
- GEP-NET: All eligible participants with Gastroenteropancreatic neuroendocrine tumor (GEP-NET) received at least one dose of Lutathera (7.4 GBq/200 mCi x 4 administrations every 8+/-1 weeks; cumulative dose: 29.6 GBq/800 mCi), with a concomitant administration of 2.5% Lysine - Arginine amino acid solution.
- PPGL: All eligible participants with Pheochromocytoma and paraganglioma (PPGL) received at least one dose of Lutathera (7.4 GBq/200 mCi x 4 administrations every 8+/-1 weeks; cumulative dose: 29.6 GBq/800 mCi), with a concomitant administration of 2.5% Lysine - Arginine amino acid solution.
Period: Overall Study
Arm/Group | GEP-NET | PPGL
Started | 4 | 7
Ongoing treatment | 0 | 1
Entered short term follow-up | 4 | 5
Entered long term follow-up | 1 | 3
Completed (Completed = Completed treatment plan) | 4 | 5
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Ongoing treatment | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The FAS included all participants that received at least one dose of Lutathera.
Groups:
- Total: Total of all reporting groups
Arm/Group | GEP-NET | PPGL | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (0.58) | 14.9 (1.77) | 15.1 (1.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 2 | 3 | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 2 | 3 | 5
  Black or African American | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Not Reported | 1 | 2 | 3
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Absorbed Radiation Doses in Target Organ
Description: Absorbed radiation doses in target organ (e.g. kidney and bone marrow) was evaluated when all Gastroenteropancreatic Neuroendocrine Tumors (GEP-NETs) and Pheochromocytoma and paraganglioma (PPGLs) as a pooled cohort patients had completed the 1st treatment of Lutathera and completed the dosimetry assessment.
Time Frame: Up to 8 days after the first Lutetium [Lu 177] dotatate dose
Population: Dosimetry Analysis Set (DAS): The DAS consisted of all participants who had at least one valid (i.e., not flagged for exclusion by the dosimetrist) dosimetry measurement.
Measure: Mean (Standard Deviation); unit: Gy/GBq
Arm/Group | GEP-NET | PPGL
Number analyzed (Participants) | 4 | 6
Gy/GBq
  Kidney | 0.71 (0.25) | 0.82 (0.32)
  Pituitary: number analyzed (Participants) | 3 | 6
  Pituitary | 1.2 (0.43) | 1.0 (0.45)
  Red Marrow (Blood) | 0.024 (0.0035) | 0.028 (0.0052)
  Red Marrow (Image) | 0.043 (0.018) | 0.067 (0.028)
  Spleen | 0.63 (0.39) | 0.82 (0.17)
  Urinary Bladder Wall | 0.50 (0.034) | 0.59 (0.096)
  Total Body | 0.040 (0.013) | 0.041 (0.0073)

2. Primary Outcome: Incidence of Adverse Events (AEs) and Lab Toxicities After 1st Lutathera Administration
Description: Safety in adolescents with SSTR-positive GEP-NETs and PPGLs as a pooled cohort was evaluated through the incidence of AEs and laboratory abnormalities after the first Lutathera dose.
Time Frame: during first cycle of Lutetium [Lu 177] dotatate treatment (Cycle = 56 days)
Population: Safety Set: The Safety Set included all participants that received at least one dose of Lutathera.
Measure: Count of Participants; unit: Participants
Arm/Group | GEP-NET | PPGL
Number analyzed (Participants) | 4 | 7
Participants | 4 | 6

3. Secondary Outcome: Incidence of Adverse Events (AEs) During Treatment and Short-term Follow-up
Description: Cumulative safety of Lutathera in adolescents with SSTR-positive GEP-NETs and PPGLs as a pooled cohort was assessed through the incidence of adverse events (AEs) and laboratory toxicities until 6 months after the last Lutathera dose.
Time Frame: From first Lutetium [Lu 177] dotatate dose to 6 months after last dose, approx. 12 months
Population: Safety Set: The Safety Set included all participants that received at least one dose of Lutathera.
Measure: Count of Participants; unit: Participants
Arm/Group | GEP-NET | PPGL
Number analyzed (Participants) | 4 | 7
Participants
  AEs during Lutathera treatment | 4 | 7
  AEs during short-term follow-up | 1 | 3

4. Secondary Outcome: Incidence of Adverse Events (AEs) During the Long Term Follow-up
Description: Long-term safety of Lutathera in adolescents with SSTR-positive GEP-NETs and PPGLs as a pooled cohort was evaluated through the incidence of AEs and laboratory abnormalities during the 5-year follow-up after the last Lutathera dose.
Time Frame: Up to 5 years after the last Lutetium [Lu 177] dotatate dose
Reporting Status: Not Posted, anticipated posting 2030-05

5. Secondary Outcome: Calculated Probability of Exceeding the Kidney and Bone Marrow External Beam Radiation Therapy (EBRT) Threshold
Description: A comparative assessment of dosimetry for organs at risk specifically kidneys and bone marrow, was performed between adolescent patients with GEP-NETs and PPGLs as a pooled cohort and adult patients using the extrapolation model developed for the clinical study to confirm the probability of exceeding 29 Gy (kidneys) & 2 Gy (bone marrow) thresholds.
Time Frame: After 4 cycles of 7.4 GBq/200 mCi; each cycle is 8+/-1 weeks
Population: Dosimetry Analysis Set (DAS) consisted of all participants who had at least one valid dosimetry measurement. Original NETTER-P protocol intended to conduct separate analyses for the GEP-NET and the PPGL populations. However, the protocol was amended to allow combined analyses for dosimetry across the two patient indications. The number of patients was equal 10, since data from one patient was excluded from the dosimetry modeling analysis, due to technical issues during image acquisitions.
Measure: Number; unit: probability
Groups:
- GEP-NET and PPGL: All eligible participants with Gastroenteropancreatic neuroendocrine tumor (GEP-NET) and Pheochromocytoma and paraganglioma (PPGL) received at least one dose of Lutathera (7.4 GBq/200 mCi x 4 administrations every 8+/-1 weeks; cumulative dose: 29.6 GBq/800 mCi), with a concomitant administration of 2.5% Lysine - Arginine amino acid solution.
Arm/Group | GEP-NET and PPGL
Number analyzed (Participants) | 10
probability
  Observed: Kidney (Probability (%) >29 Gy) | 20.0
  Observed: Bone Marrow (Probability (%) >2 Gy) | 0.0

6. Secondary Outcome: Pharmacokinetics (PK) Parameter: AUClast - Based on Blood Radioactivity Concentration Data
Description: A comparative assessment of PK will be performed between Observed and Predicted adolescent patients with GEP-NETs and PPGLs as a pooled cohort and adult patients using the extrapolation model developed for the clinical study. The observed PK metrics were calculated using non-compartmental analysis (NCA), the predicted PK metrics were derived based on the adolescent population pharmacokinetics (popPK) model.
Time Frame: Up to 72 hours after the first Lutetium [Lu 177] dotatate dose
Population: The PK Analysis Set (PKAS) consisted of all participants who had at least one valid (i.e., not flagged for exclusion) PK measurement. Original NETTER-P protocol intended to conduct separate analyses for the GEP-NET and the PPGL populations. However, the protocol was amended to allow combined analyses for PK across the two patient indications.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | GEP-NET and PPGL
Number analyzed (Participants) | 11
ng.h/mL
  Observed | 41 (24.15)
  Predicted | 32.34 (10.43)

7. Secondary Outcome: Pharmacokinetics (PK) Parameter: Cmax - Based on Blood Radioactivity Concentration Data
Description: as for outcome 6
Time Frame: Up to 72 hours after the first Lutetium [Lu 177] dotatate dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GEP-NET and PPGL
Number analyzed (Participants) | 11
ng/mL
  Observed | 11.17 (33.04)
  Predicted | 10.31 (5.22)

8. Secondary Outcome: Pharmacokinetics (PK) Parameter: Tmax - Based on Blood Radioactivity Concentration Data
Description: as for outcome 6
Time Frame: Up to 72 hours after the first Lutetium [Lu 177] dotatate dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hr
Arm/Group | GEP-NET and PPGL
Number analyzed (Participants) | 11
hr
  Observed | 0.58 [0.5 to 0.77]
  Predicted | 0.5 [0.5 to 0.7]

ADVERSE EVENTS:
Time Frame: AEs & on-treatment deaths were collected from the first dose of study treatment up to data cut-off date of 12-Mar-2024, approx. 19 months from the FPFV.
Description: Any sign or symptom that occurs during the conduct of the trial.
Groups:
- Total: All participants from the GEP-NET and PPGL arms.
Arm/Group | GEP-NET | PPGL | Total
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/7 | 2/11
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GEP-NET (N=4) | PPGL (N=7) | Total (N=11)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GEP-NET (N=4) | PPGL (N=7) | Total (N=11)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 3
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1
Photophobia (Eye disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 3
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 4
Vomiting (Gastrointestinal disorders) | 1 | 2 | 3
Asthenia (General disorders and administration site conditions) | 1 | 0 | 1
Fatigue (General disorders and administration site conditions) | 1 | 2 | 3
Influenza like illness (General disorders and administration site conditions) | 1 | 1 | 2
Pyrexia (General disorders and administration site conditions) | 0 | 1 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Otitis media (Infections and infestations) | 0 | 1 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 1
Tinea versicolour (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 2
Viral infection (Infections and infestations) | 1 | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 2 | 2
Lymphocyte count decreased (Investigations) | 0 | 3 | 3
Neutrophil count decreased (Investigations) | 0 | 2 | 2
Weight decreased (Investigations) | 1 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 2 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 2
Headache (Nervous system disorders) | 2 | 4 | 6
Hypersomnia (Nervous system disorders) | 1 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1
Phonophobia (Psychiatric disorders) | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Hot flush (Vascular disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e., data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT04711135/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT04711135/SAP_001.pdf